CLINICAL TRIAL: NCT05227248
Title: Evaluation of the Effects of Chocolate on Anatomy and Functionality of Retinal Blood Vessels
Brief Title: Chocolate Dynamic Vessel Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Querques Giuseppe (Other)
Responsible Party: Sponsor-Investigator, Querques Giuseppe, Professor, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: FondazioneSanRaffaele
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Retinal Vascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main study arm (Experimental): Patients received intervention 1 and then intervention 2 after 7 weeks
  Interventions: Dietary Supplement: Dark chocolate; Dietary Supplement: Milk Chocolate

INTERVENTIONS:
Dietary Supplement: Dark chocolate — Patients were administered 20 grams of dark chocolate
Dietary Supplement: Milk Chocolate — Patients were administered 7.5 grams of milk chocolate

SUMMARY:
The study aims at evaluating the effect of dark chocolate consumption on anatomy and functionality of retinal blood vessels by comparing these same parameters after milk chocolate consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Healthy volunteers
* No vascular diseases
* No ocular diseases
* Volunteers capable of understanding informed consent

Exclusion Criteria:

* Patient unable to follow the instructions
* Patient unable to come back for follow-up
* opacity of lens, cornea, or vitreous
* Allergies that contraindicate pupil dilation
* Eye diseases
* Myopia greater than -8.0 Diopter (D),
* Hyperopia greater than 5.0 D
* Astigmatism greater than -3.0 D

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Retinal perfusion | Baseline, 2 hours after intervention
  Changes in retinal perfusion using Optical Coherence Tomography Angiography
Retinal vascular response | Baseline, 2 hours after intervention
  Changes in retinal vascular response to flicker stimulation using Dynamic Vessels Analysis and Retinal Vessels Analysis

SECONDARY OUTCOMES:
Visual Acuity | Baseline, 2 hours after intervention
  Best Corrected Visual Acuity changes

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandello, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Giuseppe Querques, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Carlo TE, Romano A, Waheed NK, Duker JS. A review of optical coherence tomography angiography (OCTA). Int J Retina Vitreous. 2015 Apr 15;1:5. doi: 10.1186/s40942-015-0005-8. eCollection 2015. PMID 27847598
- [Background] Huang Y, Zhang Q, Thorell MR, An L, Durbin MK, Laron M, Sharma U, Gregori G, Rosenfeld PJ, Wang RK. Swept-source OCT angiography of the retinal vasculature using intensity differentiation-based optical microangiography algorithms. Ophthalmic Surg Lasers Imaging Retina. 2014 Sep-Oct;45(5):382-9. doi: 10.3928/23258160-20140909-08. PMID 25230403
- [Background] McClintic SM, Jia Y, Huang D, Bailey ST. Optical coherence tomographic angiography of choroidal neovascularization associated with central serous chorioretinopathy. JAMA Ophthalmol. 2015 Oct;133(10):1212-4. doi: 10.1001/jamaophthalmol.2015.2126. No abstract available. PMID 26135638
- [Background] Siedlecki J, Mohr N, Luft N, Schworm B, Keidel L, Priglinger SG. Effects of Flavanol-Rich Dark Chocolate on Visual Function and Retinal Perfusion Measured With Optical Coherence Tomography Angiography: A Randomized Clinical Trial. JAMA Ophthalmol. 2019 Dec 1;137(12):1373-1379. doi: 10.1001/jamaophthalmol.2019.3731. PMID 31556937
- [Background] Rabin JC, Karunathilake N, Patrizi K. Effects of Milk vs Dark Chocolate Consumption on Visual Acuity and Contrast Sensitivity Within 2 Hours: A Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jun 1;136(6):678-681. doi: 10.1001/jamaophthalmol.2018.0978. PMID 29710322
- [Derived] Sacconi R, Pezzella M, Ribarich N, Menean M, Servillo A, Bandello F, Querques G. Benefits of dark chocolate intake on retinal vessels functionality: a randomized, blind, crossover clinical trial. Sci Rep. 2024 Aug 30;14(1):20203. doi: 10.1038/s41598-024-70289-7. PMID 39215063
- See also: Nutrition Foundation of Italy — https://www.nutrition-foundation.it/